CLINICAL TRIAL: NCT06027580
Title: Assessing Functional Improvements With Use of the SPIO Core-Max Expedition TLSO
Brief Title: Orthosis to Improve Trunk Control in Infants Age 6-18 Months
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: SPIO (Unknown)
Responsible Party: Principal Investigator, Mitchell O'Neill, Assistant Professor, Medical College of Wisconsin
Other Study IDs: PRO00048530
Record Dates: First submitted 2023-08-09; First posted 2023-09-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
Keywords: abnormal muscle tone; cerebral palsy; hypotonia; muscle tone; spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Hypotonia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SPIO group: Standard Care Therapy option 1: parents may self-select this standard care combined option of therapy and use of SPIO® Core-MAX® Expedition thoracolumbosacral orthosis
  Interventions: Device: SPIO® Core-MAX® Expedition thoracolumbosacral orthosis
- Control group: Standard Care Therapy option 2: parents may self-select this standard care option of therapy alone
  Interventions: Other: Standard Care Therapy option

INTERVENTIONS:
Device: SPIO® Core-MAX® Expedition thoracolumbosacral orthosis — SPIO® Core-MAX® Expedition thoracolumbosacral orthosis use 2 hours per day for 6 months
  Groups: SPIO group
Other: Standard Care Therapy option — Standard of care Therapy without the use of trunk orthosis
  Groups: Control group

SUMMARY:
The purpose of this study is to determine the impact of the SPIO® Core-MAX® Expedition orthosis on an infant's head, trunk and upper limb function.

DETAILED DESCRIPTION:
This study will observe the difference in outcomes between two courses of standard clinical care: therapy or therapy with the SPIO® Core-MAX® Expedition orthosis. Families will self-select that standard care option that works best for their family, and outcomes will be observed at baseline, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects aged 6 months to 18 months age corrected with abnormal muscle tone
* No previous use of SPIO® or similar Lycra/compression garments
* Assessed by provider as likely to benefit from use of compression garment

Exclusion Criteria:

* Non-English speaking
* Inability for family to bring study subject to assessments
* Orthosis or casting that contraindicate SPIO® Core-MAX® during the study period
* Botulinum toxin injections within 3 months, or during study participation
* Having prior orthopedic or neurosurgery surgeries within one year

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6 months to 18 months age corrected with abnormal muscle tone assessed by a provider as likely to benefit from use of a compression garment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Change in head and trunk position from centerline at baseline, 3-months and 6-months. | Through study completion, an average of 2 years
  Degree change in head and trunk position from centerline as assessed by motion capture.
Change from baseline to 3-months and 6-months on the Pediatric Quality of Life Inventory Infant Scale. | Through study completion, an average of 2 years
  The Pediatric Quality of Life Inventory Infant Scales (PedQL-I) is used to assess parent-reported health-related quality of life for children with ages 1-12 months or 12-24 months. It has the same five components, including physical functioning (6 items), physical symptoms (10 items), emotional functions (12 items), social functioning (4 items), and cognitive functioning (4 items) with scale from 0 to 4.
  0 if it is never a problem
  1. if it is almost never a problem
  2. if it is sometimes a problem
  3. if it is often a problem
  4. if it is almost always a problem

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell O'Neill, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No